CLINICAL TRIAL: NCT04222205
Title: A Cluster-Randomized Crossover Trial to Compare Spontaneous Breathing Trial With T-piece or Inspiratory Pressure Augmentation
Brief Title: Spontaneous Breathing Trial With T-piece or Inspiratory Pressure Augmentation
Acronym: SBT-TIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 201901036RINA
Record Dates: First submitted 2019-12-08; First posted 2020-01-09 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Ventilator Weaning
Keywords: Clinical trial; Mechanical ventilation; Respiratory failure; Spontaneous breathing trial; Weaning
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Serum Bactericidal Test

STUDY DESIGN:
Intervention Model Description: Cluster-Randomized Crossover Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crossover sequence 1 (Active Comparator): Cluster-randomization crossover sequence 1:
  T-piece during odd-numbered months and inspiratory pressure augmentation during even-numbered months.
  Interventions: Diagnostic Test: Spontaneous breathing trial (SBT) crossover sequence 1
- Crossover sequence 2 (Experimental): Cluster-randomization crossover sequence 2:
  T-piece during even-numbered months and inspiratory pressure augmentation during odd-numbered months.
  Interventions: Diagnostic Test: Spontaneous breathing trial (SBT) crossover sequence 2

INTERVENTIONS:
Diagnostic Test: Spontaneous breathing trial (SBT) crossover sequence 1 — SBTs with T-piece breathing for one hour during odd-numbered months and SBTs with inspiratory pressure augmentation for one hour during even-numbered months.
  Arms: Crossover sequence 1
Diagnostic Test: Spontaneous breathing trial (SBT) crossover sequence 2 — SBTs with inspiratory pressure augmentation for one hour during odd-numbered months and SBTs with T-piece breathing for one hour during even-numbered months.
  Arms: Crossover sequence 2

SUMMARY:
Weaning is an important process to gradually separate mechanically ventilated patients from ventilators. A good weaning strategy aims to early identify mechanically ventilated patients who are ready for extubation but not to prematurely extubate them. Spontaneous breathing trial (SBT) is a test to assess the patient's ability to breathe spontaneously when extubated. Several methods have been used to conduct an SBT, including T-piece breathing, low-level pressure support ventilation (PSV) of 5-7 cm H2O, continuous positive airway pressure and automatic tube compensation (ATC).

The investigators hypothesized that an SBT with inspiratory pressure augmentation increases initial SBT success, reduces the length of invasive mechanical ventilation (iMV) support and does not increase reintubation risk as compared with T-piece, which result in a higher proportion of patients successfully liberated from iMV in the inspiratory pressure augmentation group. However, inspiratory pressure augmentation significantly reduces work of breathing on an SBT as compared with T-piece. Patients extubated following an SBT with inspiratory pressure augmentation may experience increased respiratory effort after extubation and this may increase the use of noninvasive ventilation after extubation. An SBT with inspiratory pressure augmentation increases iMV free days but not MV free days as compared with T-piece. Longer iMV free days may be associated with a lower mortality due to fewer iMV related complication.

This study is a pragmatic, cluster-randomized, multiple crossover, multicenter trial to compare SBTs with T-piece versus inspiratory pressure augmentation in weaning outcomes. Mechanically ventilated patients who meet the criteria for readiness to SBT will be included. The patients will use either T-piece or inspiratory pressure augmentation as SBT for weaning according to an ICU-based cluster randomization and crossover sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the adult intensive care unit (ICU)
2. Receiving invasive mechanical ventilation via an endotracheal tube
3. Ready to start an SBT* *The criteria of readiness to an SBT include FiO2 ≤ 0.4, PEEP ≤ 8 cmH2O, minute ventilation ≤ 0.15 L/min/predicted body weight, inspiratory pressure or driving pressure ≤ 14 cm H2O, stable cardiovascular status and no worsening of non-pulmonary organ function.

Exclusion Criteria:

1. Age < 20 years
2. Receiving mechanical ventilation via tracheostomy
3. Mechanical ventilation < 12 hours
4. Invasive ventilation started before the index hospitalization
5. On do-not-intubate order

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2143 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful liberation from invasive mechanical ventilation | ICU discharge, up to 28 days after the initial SBT
  The primary study endpoint is to compare the effect of SBT with T-piece versus inspiratory pressure augmentation on the proportion of patients with successful liberation from invasive mechanical ventilation in the ICU among patients who have started an SBT. Successful liberation is defined as sustaining iMV free for at least five days after extubation.

SECONDARY OUTCOMES:
Successful liberation from invasive and noninvasive mechanical ventilation | ICU discharge, up to 28 days after the initial SBT
  Proportion of successful liberation from invasive and noninvasive mechanical ventilation in the ICU.
Successful liberation from invasive mechanical ventilation | 28 days
  Proportion of successful liberation from invasive mechanical ventilation on day 28 from intubation.
Time to successful liberation from invasive mechanical ventilation | 28 days
  Time to successful liberation from invasive mechanical ventilation using competing-risks analysis.
Time to successful liberation from invasive and noninvasive mechanical ventilation | 28 days
  Time to successful liberation from invasive and noninvasive mechanical ventilation using competing-risks analysis.
Intubation free days | 28 days
  The number of days that a patient is alive and free from intubation.
Adjusted risk ratio of successful liberation from invasive mechanical ventilation | ICU discharge, up to 28 days after the initial SBT
  Adjusted risk ratio of successful liberation from invasive mechanical ventilation for T-piece versus inspiratory pressure augmentation group.
Initial SBT success | During the ICU stay, up to 28 days
  Proportion of initial SBT success among patients who have started an SBT.
Extubation failure | Five days from extubation
  Proportion of extubation failure among patients undergoing planned extubation.
Proportion of planned extubation | ICU discharge, up to 28 days after the initial SBT
  Proportion of planned extubation in the ICU
Use of noninvasive ventilation after extubation | Five days from extubation
  Proportion of use of noninvasive ventilation (>24 hours) after extubation.
ICU mortality | ICU discharge, up to 28 days after the initial SBT
  Proportion of death in the ICU.
28-day mortality | 28 days
  Probability of death in 28 days using kaplan-meier estimator.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fu-Chang Tsai, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei, Please Select
  - National Taiwan University Hospital Hsin-Chu Branch, Taoyuan District
  - National Taiwan University Hospital Yunlin Branch, Yunlin

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data are available from the corresponding author on reasonable request.